CLINICAL TRIAL: NCT06301763
Title: Oral Enteral Nutrition in Delayed Onset Radiotherapy-related Swallowing Disorder in Nasopharyngeal Carcinoma: A Randomly Controlled Study
Brief Title: Oral Enteral Nutrition in Delayed Onset Radiotherapy-related Swallowing Disorder in Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nosencekCancer-old
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oral-esophageal Tube Feeding (Experimental): During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on health condition. The observation group receives IOE for enteral nutrition support.54 cm.
  Interventions: Device: Intermittent Oral-esophageal Tube Feeding
- nasogastric tube feeding (Active Comparator): During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on health condition.The control group receives NGT for enteral nutrition support
  Interventions: Device: nasogastric tube feeding

INTERVENTIONS:
Device: Intermittent Oral-esophageal Tube Feeding — During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on the health condition.The observation group receives Intermittent Oral-esophageal Tube Feeding for enteral nutrition support (developed by the Dysphagia Institute of Zhengzhou University, CN201821314797.2), which is made of silicone material, 40 cm long, with an inner diameter of 0.54 cm.
  Arms: Intermittent Oral-esophageal Tube Feeding
Device: nasogastric tube feeding — During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on the health condition.The control group is provided with nutritional support as nasogastric tube feeding, performed 6-10 times per day according to relevant guidelines, with an interval of more than 2 hours between every two feedings, and a feeding volume not exceeding 200 ml per time.
  Arms: nasogastric tube feeding

SUMMARY:
This is a prospective multicenter study with patients with delayed dysphagia after radiotherapy for NPC. Patients enrolled are randomly divided equally into the observation group and the control group. All patients receive conventional care, and the observation group received IOE while the control group received NGT for enteral nutrition support. Baseline information (demographics, medical history, etc.), nutritional status at admission and after treatment, depression, dysphagia, and quality of life (QOL) after treatment as well as adverse events are compared.

DETAILED DESCRIPTION:
Palliation to delayed dysphagia after radiotherapy for nasopharyngeal carcinoma (NPC) continues to be a challenge. Although nasogastric tube feeding (NGT) has been adopted widely, the weaknesses have yet to be improved by another enteral nutrition support mode. This study aims to observe the clinical efficacy of intermittent oro-esophageal tube feeding (IOE) in the treatment of delayed dysphagia after radiotherapy for (NPC). This is a prospective multicenter study with patients with delayed dysphagia after radiotherapy for NPC. Patients enrolled are randomly divided equally into the observation group and the control group. All patients receive conventional care, and the observation group received IOE while the control group received NGT for enteral nutrition support. Baseline information (demographics, medical history, etc.), nutritional status at admission and after treatment, depression, dysphagia, and quality of life (QOL) after treatment as well as adverse events are compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* With the history of Nasopharyngeal Carcinoma and radiation therapy.
* With dysphagia occurred at least three years after radiotherapy (confirmed by videofluoroscopic swallowing study), in need of and feasible for enteral nutrition support.
* Conscious and with stable vital signs;
* Willing to participate and sign the written informed consent form either personally or by a family member.

Exclusion Criteria:

* Presence of other diseases that might cause dysphagia.
* With distant metastasis of tumors, or complicated with severe systemic disorders or malignancies.
* Concurrent participation in other treatments that could interfere with the trial.
* Inability to cooperate with treatment due to aphasia, mental health issues, etc.
* Received tube feeding for enteral nutrition support within the past three years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin Level | day 1 and day 15
  Hemoglobin was recorded through the blood routine test. (Hb, g/L)
Serum albumin Level | day 1 and day 15
  Serum albumin was recorded through the blood routine test. (ALB, g/L)
Total serum protein Level | day 1 and day 15
  Total serum protein was recorded through the blood routine test. (TP, g/L)
Serum prealbumin Level | day 1 and day 15
  Serum prealbumin was recorded through the blood routine test.(PA, g/L)
Body Mass Index Level | day 1 and day 15
  Body Mass Index was assessed with the combination of body weight and height: weight (kg)/ [height (m)] ^2

SECONDARY OUTCOMES:
Depression | day 1 and day 15
  The PATIENT HEALTH QUESTIONNAIRE scale is utilized to evaluate the depression of patients at admission and after treatment. Options representing varying degrees of severity, ranging from 0 to 3 were provided in each aspect. The total scores between 0 and 4 were classified as negative, indicating the absence of depressive symptoms, while scores above 4 were classified as positive, indicating the presence of potential depressive symptoms.
Swallowing-Quality of Life questionnaire | day 1 and day 15
  The Chinese version of the Swallowing-Quality of Life questionnaire (SWAL-QOL) was used to assess the quality of life of patients.he Likert scale ranging from 1 to 5 was utilized for scoring, with a total of 44 items, including difficulties in swallowing, dietary restrictions, oral health, social communication, and others. The total score was converted to a standard percentage scale ranging from 0 to 100, with positively correlated with QOL.
Functional Oral Intake Scale | day 1 and day 15
  The Functional Oral Intake Scale (FOIS) was used to evaluate function of oral intake. In the FOIS assessment, two professional rehabilitation therapists communicated with the patients, observed and recorded to assess their swallowing function. The assessment scale consists of seven levels, with a higher level indicating progressively better swallowing function (less dysphagia).
Penetration-Aspiration Scale | day 1 and day 15
  In this study, the Penetration-Aspiration Scale (PAS) was recruited, which was a commonly used to evaluate the occurrence of penetration or aspiration during swallowing. It categorizes dysphagia into eight levels, with Level 0 indicating no penetration or aspiration and Level 8 indicating severe aspiration. A higher level indicates more severe dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group
Locations (1):
- Afli Hospital, Zhongguo, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng H, Zhao W, Zhang X, Wang X, Luo P, Li H, Wang L, Zeng X. How enteral nutrition modes influence nasopharyngeal carcinoma survivors with late dysphagia after radiotherapy: a randomized controlled study. Support Care Cancer. 2024 Oct 5;32(10):702. doi: 10.1007/s00520-024-08912-6. PMID 39367230